CLINICAL TRIAL: NCT01720303
Title: A Multi-centre, Open, Randomised, Parallel, Controlled Trial to Compare the Efficacy and Safety of Repaglinide Combined With Bedtime Insulin With Insulin Alone in Type 2 Diabetic Subjects Inadequately Controlled With Sulphonylurea ± Biguanide Therapy
Brief Title: Efficacy and Safety of Repaglinide Combined With Insulin in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-3020
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Insulin, Isophane; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rep + NPH (Experimental)
  Interventions: Drug: repaglinide; Drug: isophane human insulin
- Premixed insulin/NPH (Active Comparator)
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: repaglinide — 2 mg (tablets) before each main meal
  Arms: Rep + NPH
Drug: isophane human insulin — Injection s.c. (under the skin) at bedtime
  Arms: Rep + NPH
Drug: insulin — Injection s.c. (under the skin) twice daily
  Arms: Premixed insulin/NPH

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare oral anti-diabetic drug (OAD) combined with insulin vs. insulin alone in subjects with type 2 diabetes not adequately controlled on the current OAD therapy.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 7.5 % and 13.0% (both inclusive)
* Fasting C-peptide above or equal to 0.33 nmol/l
* BMI (Body Mass Index) between 25 and 32 kg/m2 (both inclusive)

Exclusion Criteria:

* Medical history of treatment with insulin within the last 6 months
* Impaired renal function, defined as serum creatinine above to 1.7 mg/dl (150 µmol/l)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2002-09-19 (Actual); Primary Completion 2003-04-10 (Actual); Study Completion 2003-04-10 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c

SECONDARY OUTCOMES:
Change in FBG (Fasting Blood Glucose)
Change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- China (2):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com